CLINICAL TRIAL: NCT06901570
Title: Clinical Assessment of Aromatic Wentong for Coronary Microvascular Disease Management
Brief Title: Clinical Evaluation of Aromatic Wentong in the Treatment of Coronary Microvascular Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xianlun Li, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023ZD0505705
Record Dates: First submitted 2025-03-11; First posted 2025-03-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Drug: Kuangxiong Aerosol
- Control Arm (Placebo Comparator)
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Kuangxiong Aerosol — Patients in the intervention group will receive Kuangxiong Aerosol for eight weeks, in addition to guideline-recommended medications. The aerosol will be administered sublingually (under the tongue), with a dosage of two sprays per dose, three times daily.
  Arms: Experimental Arm
Drug: Placebo Drug — Patients in the control group will receive a placebo version of Kuangxiong Aerosol for eight weeks, alongside guideline-recommended medications. The placebo will be administered sublingually (under the tongue), with a dosage of two sprays per dose, three times daily.
  Arms: Control Arm

SUMMARY:
Coronary Microvascular Disease (CMD) is a condition where patients experience chest pain (angina) even though their coronary arteries appear normal on angiography. It is common among people with coronary heart disease, especially those with chest pain as their main symptom. Unfortunately, there are no effective treatments available for these patients, and symptoms like chest tightness and persistent pain greatly affect their quality of life.

Traditional Chinese Medicine (TCM) suggests that the root cause of microvascular disease is blocked collateral blood vessels. Aromatic Wentong, a TCM approach, aims to improve blood flow and relieve blockages. Kuangxiong Aerosol is a Chinese patent medicine developed based on the principles of Aromatic Wentong.

This study is a multicenter, randomized, double-blind, placebo-controlled trial involving 528 patients with chest pain and suspected CMD. Participants are recruited from several hospitals, including China-Japan Friendship Hospital, Fuwai Hospital, and Xiyuan Hospital. Patients are randomly divided into two groups:

The intervention group receives standard guideline-recommended treatment plus Kuangxiong Aerosol.

The control group receives standard treatment plus a placebo version of Kuangxiong Aerosol.

The treatment lasts for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years, regardless of gender.
* Clinical symptoms of myocardial ischemia.
* Objective evidence of myocardial ischemia, including:

  1. ECG changes during chest pain episodes,
  2. Stress test-induced chest pain symptoms and/or abnormal myocardial blood flow and/or abnormal cardiac wall motion with ischemic ECG changes.
* Coronary angiography (CAG) showing >50% reduction in the diameter of the epicardial coronary artery.
* QFR > 0.80 and AMR > 2.5 mmHg·s/cm.
* Discontinuation of all Chinese medicine interventions for at least two weeks prior to enrollment.
* Provision of informed consent and a signed informed consent form.

Exclusion Criteria:

* Significant liver or kidney dysfunction, defined as ALT, AST, or blood creatinine levels >3 times the upper limit of normal.
* Severe cardiac conditions, including heart failure, myocarditis, cardiomyopathy, acute pericarditis, structural heart disease.
* Severe systemic diseases, such as severe mental illness, hematopoietic system disorders, or malignant tumors.
* Suspected or confirmed allergy to the trial drug.
* Individuals deemed by researchers to be unsuitable for participation in the clinical trial.
* Women who are pregnant, planning to become pregnant, or currently lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Score of the Seattle Angina Questionnaire | Baseline, 4 weeks, and 8 weeks
  The Seattle Angina Questionnaire (SAQ) is a 19-item self-administered, disease-specific patient-reported outcome with 5 domains: physical limitation (Question 1), anginal stability (Question 2), anginal frequency (Question 3), treatment satisfaction (Question 4-8), and disease perception/quality of life (Question 9-11). All SAQ domain scores and the summary score range from 0 to 100 with higher scores indicating less angina, fewer functional limitations, and better quality of life.

SECONDARY OUTCOMES:
Score of the Traditional Chinese Medicine Syndrome Score Scale | Baseline, 4 weeks, and 8 weeks.
  The Traditional Chinese Medicine Syndrome Score Scale is a scale based on patients' syndromes and signs, and it varies depending on the disease and context. In this study, the Traditional Chinese Medicine Syndrome Score Scale consists of 14 items, each scored from 0 to 4. The sum of all items represents the final score, where a higher score indicates worse symptoms and a lower score indicates better symptoms.
Score of the Medical Outcomes Study 36-Item Short-Form Health Survey | Baseline, 4 weeks, and 8 weeks
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) includes eight scaled scores: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The scores are weighted sums of the questions in each section. Scores range from 0 to 100, where lower scores indicate more disability and higher scores indicate less disability.
Levels of inflammatory factors (CRP, hs-CRP, IL-1β, IL-6) | Baseline, 8 weeks
Levels of vascular endothelial function markers (NO, ET-1) | Baseline, 8 weeks
Factors and levels of transcriptomics | Baseline, 8 weeks
Factors and levels of proteomics | Baseline, 8 weeks
Factors and levels of metabolomics | Baseline, 8 weeks
Myocardial contrast echocardiography | Baseline, 8 weeks
  A subset of 40 patients from each group will undergo myocardial contrast echocardiography to assess myocardial blood flow and coronary flow reserve.
Major adverse cardiovascular events | 8 weeks
  The major adverse cardiovascular events are defined by the combination of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, rehospitalization for heart failure, or unstable angina pectoris.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Chaoyang District, China

IPD SHARING:
Plan to Share IPD: No